CLINICAL TRIAL: NCT05030363
Title: The Efficacy and Safety of Alcoholic Dehydrogenase (ALDH) Enzyme Supplement in Chemotherapy-Related Fatigue With Advanced Gastrointestinal Cancer Patients: A 2-Period, Crossover, Single-Center Study
Brief Title: ALDH Enzyme in CRF With Advanced GI Cancer
Acronym: ALDHCRF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: PicoEnTech001
Record Dates: First submitted 2021-08-09; First posted 2021-09-01 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Fatigue; Gastrointestinal Cancer; Aldehyde Dehydrogenase
Keywords: Chemotherapy-Related Fatigue; Gastrointestinal Cancer; Aldehyde Dehydrogenase
MeSH Terms: conditions — Fatigue; Gastrointestinal Neoplasms

STUDY DESIGN:
Intervention Model Description: A 2-Period, Crossover, Single-Center Study
Masking Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Upfront ALDH enzyme supplement (Experimental): Upfront ALDH enzyme supplement; After randomization, patients will receive ALDH enzyme supplement twice a day for consecutive 14 days during chemotherapy (period 1; day 1 to day 14) until unacceptable toxicity, or consent withdrawal. Patients will visit clinic on day 15, then will be followed on day 29 without ALDH enzyme administration during subsequent chemotherapy (period 2).
  Interventions: Drug: ALDH enzyme supplementation
- Delayed ALDH enzyme supplement (Other): Delayed ALDH enzyme supplement; patients will not take ALDH enzyme supplement during chemotherapy after randomization on day 1 to day 14 (period 1). On day 15, Patients will visit for subsequent chemotherapy and start ALDH enzyme supplement twice a day for 14 consecutive days during chemotherapy (period 2; day 15 to day 29).
  Interventions: Drug: ALDH enzyme supplementation

INTERVENTIONS:
Drug: ALDH enzyme supplementation — ALDH enzyme (PICOZYMEQ™)

SUMMARY:
Aldehyde dehydrogenase (ALDH) enzyme supplementation plays an essential role in the elimination of toxic metabolites and reduction of reactive oxygen species bioactivation, which can protect and relieve chemotherapy-related fatigue (CRF) in cancer patients. The aim of this study is to evaluate the efficacy and safety of ALDH enzyme in CRF with advanced gastrointestinal cancer patients. The primary endpoint is the change of FACIT-F (Functional Assessment of Chronic Illness Therapy-Fatigue) score on day 15 compared to baseline after chemotherapy. The secondary endpoint including change of FACIT-F on day 29 compared to day 15, change of ESAS (Edmonton Symptom Assessment System) on day 15 compared to baseline, safety and toxicities, and exploratory biomarkers.

DETAILED DESCRIPTION:
Chemotherapy-related fatigue (CRF) occurs universally in cancer patients which can be a debilitating symptom that affects patients' quality of life. The impact of CRF has been associated with mood disorder, sleep disturbance, cognitive dysfunction, inflammation mediated putative biological disturbances, and functional morbidities. Although the etiology is heterogeneous and complex, one of the proposed mechanisms is that chemotherapy induced multiple oxidative degradation of the lipid membrane which generates reactive oxygen species (ROS) and tissue damage. These conditions result in inflammation-induced reduction in central dopaminergic neurotransmission, nutritional deficiency (especially in vitamins and minerals), and immunodeficiency, which clinically manifest as CRF. To date, various agents including psychostimulants (methylphenidate, donepezil, and modafinil), dexamethasone, and Korean red ginseng (KRG) were used in the management of CRF. However, the prevalence of CRF is still high primarily due to lack of proven effective therapies. ALDH enzyme supplementation plays an essential role in the eliminates 4-hydoxynonenal, malondialdehyde from lipid peroxidation and reduce ROS bioactivation, which can protect and relieve CRF in cancer patients. Based on these rational backgrounds, the aim or this study is to evaluate the efficacy and safety of ALDH enzyme in CRF with advanced gastrointestinal cancer patients.

ELIGIBILITY:
Inclusion Criteria:

To be included in the trial, subjects must meet all of the following criteria:

1. Fatigue score ≥ 4 on analog scale of 0 to 10 (0; not at all, 10; worst possible fatigue) for more than 1 week.
2. Subject has willing and able to written informed consent form (ICF) prior to any screening procedures.
3. Age ≥ 19 years old of male and female.
4. Life expectancy more than 3 months.

Exclusion Criteria:

1. Hb < 8g/dL
2. Uncontrolled hyper- or hypothyroidism despite of appropriate treatment
3. Evidence of central nervous system (CNS) tumor metastasis; permitted if asymptomatic or neurologically stable.
4. Sign of active and uncontrolled bacterial or viral infection requiring systemic therapy
5. Abnormal cognition status or psychiatric disease.
6. Anamnesis of hypersensitivity reaction to the ALDH enzyme.
7. Current use or previous use within 14 days of the following medications: Korean-Chinese medications, methylphenidate, modafinil, phenobarbital, diphenylhydantoin, primidone, phenylbutazone, monoamine oxidase inhibitors, clonidine, and tricyclic antidepressants.
8. Medical conditions that could affect trial outcomes or subjects who were considered unsuitable for trial enrollment by the investigator.

Ages: 19 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2021-10-25 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of FACIT-F score | Day 15 compared to baseline
  Change of FACIT-F score on day 15 compared to baseline after chemotherapy

SECONDARY OUTCOMES:
Change of FACIT-F score | Day 29 compared to day 15
  Change of FACIT-F score on day 29 compared to day 15 after chemotherapy
Change of ESAS | Day 15 compared to baseline
  Change of ESAS on day 15 compared to baseline after chemotherapy
Change of ESAS | Day 29 compared to day 15
  Change of ESAS on day 29 compared to day 15 after chemotherapy
Incidence of treatment-related adverse events | Day 15 and 29
  Safety and tolerability assessments
Exploratory biomarker studies - Urine malondialdehyde - ALDH2 polymorphism (ALDH2 *1/*2, rs671 A/G) - Change of inflammatory cytokines | Day 1, 15 and 29
  Analysis Inflammatory cytokine and metabolites during ALDH enzyme supplement and explore predictive biomarker using urine malondialdehyde

CONTACTS AND LOCATIONS:
Overall Officials: Soohyeon Lee, MD, PhD, Principal Investigator — Korea University Anam Hospital
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No